CLINICAL TRIAL: NCT05033964
Title: The DESyne BDS Plus RCT: A Randomized Clinical Trial to Assess the Elixir DESyne BDS Plus Drug Eluting Coronary Stent System for the Treatment of de Novo Native Coronary Artery Lesions
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELX-CL-2005
Record Dates: First submitted 2021-08-17; First posted 2021-09-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Coronary Stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: prospective, multi-center, single blind, randomized clinical study. Randomization is 1:1
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- DESyne BDS Plus Arm (Experimental): DESyne BDS Plus Drug Eluting Coronary Stent System (DESyne BDS Plus DECSS; DESyne BDS Plus) is loaded with Sirolimus, Rivaroxaban and Argatroban
  Interventions: Combination Product: Percutaneous Coronary Intervention with drug eluting stents
- DESyne X2 Arm (Active Comparator): The DESyne X2 Novolimus Eluting Coronary Stent System (DESyne X2 NECSS; DESyne X2) is loaded with Novolimus
  Interventions: Combination Product: Percutaneous Coronary Intervention with drug eluting stents

INTERVENTIONS:
Combination Product: Percutaneous Coronary Intervention with drug eluting stents — Coronary drug eluting stent implantation

SUMMARY:
The objective of this clinical trial is to confirm the safety, effectiveness and performance of the DESyne BDS Plus Drug Eluting Coronary Stent System (DESyne BDS Plus DECSS) (Test) as compared to the CE Mark approved DESyne X2 Novolimus Eluting Coronary Stent System (DESyne X2 NECSS; DESyne X2) (Control) in the treatment of de novo native coronary artery lesions.

DETAILED DESCRIPTION:
The DESyne BDS Plus Randomized Clinical Trial is a prospective, multi-center, single blind, randomized clinical study. Randomization (1:1; DESyne BDS Plus : DESyne X2) of up to 200 patients (100 in each arm) requiring treatment of up to two de novo coronary artery lesions ≤ 34 mm in length in vessels ≥ 2.25 mm and ≤ 3.5 mm in diameter will be conducted. The study will be conducted in two parts, with randomization of the first 100 subjects (Cohort 1) followed by the randomization of an additional 100 subjects (Cohort 2).

In an imaging subset of approximately 60 subjects (30 per arm), Angiography and OCT will be performed at index procedure, and again at 6-month follow-up.

The PK sub-study will enroll up to 10 non-randomized subjects treated only with the DESyne BDS Plus device, with a maximum of three DESyne BDS Plus stents implanted. The PK sub-study is being conducted to assess the blood pharmacokinetics of the three drugs (Sirolimus, Rivaroxaban, Argatroban) eluted from the DESyne BDS Plus after implantation. PK measurements will be conducted at 10 minutes, 30 minutes, 1, 2, 4, 6, 12, 24, 72 hours, and 7 days. In addition, all PK subjects will undergo clinical assessments/follow-up at 3 days or hospital discharge (whichever comes first), 1 month, 6 months, 12 months, 2 years, and 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age
2. Patient is able to understand the risks, benefits and treatment alternatives of receiving the DESyne BDS Plus DECSS or the DESyne X2 NECSS and provide written informed consent or oral consent (in urgent PCI) as allowed per hospital standard and as approved by the local Ethics Committee, prior to any clinical study-related procedure
3. Indication for a percutaneous intervention with stent implantation in native epicardial arteries including patients with stable coronary artery disease and acute coronary syndromes including NSTEMI and STEMI.
4. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
5. Patient agrees to undergo all clinical study required follow up visits, angiograms, and imaging testing (as applicable)
6. Patient agrees not to participate in any other clinical research study for a period of one year following the index procedure (long term follow-up or observational studies are permitted)

   Angiographic Inclusion Criteria
7. Target lesion(s) must be de novo coronary artery lesion(s) and must be located in a separate* vessel from other target or non-target lesions.
8. Target lesion(s) must have a reference vessel diameter (RVD) of ≥ 2.25 and ≤ 3.5 mm by visual estimation
9. Target lesion(s) must measure ≤ 34 mm in length, and able to be covered by a single device with 2 mm of healthy vessel on either side of planned implantation site
10. Target lesion(s) must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and <100%. When two target lesions are treated, they must be located in separate major epicardial vessels

    Additional Inclusion Criteria for PK study:
11. Patients participating in PK study must meet all general and angiographic inclusion/exclusion criteria and may be treated with only the DESyne BDS Plus during Index Procedure.

Exclusion Criteria:

1. Acute myocardial infarction with Killip Class III and IV
2. Acute myocardial infarction requiring resuscitation
3. Acute myocardial infarction requiring IABP or ventilation support
4. Patient had fibrinolysis prior to PCI
5. Patient has current unstable ventricular arrhythmias
6. Patient has a known left ventricular ejection fraction (LVEF) < 30%
7. Patient has received a heart transplant or any other organ transplant or is on a waiting list for an organ transplant
8. Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
9. Patient is receiving immunosuppression therapy, other than steroids or has known immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.)
10. Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, prasugrel or ticagrelor, Novolimus, Sirolimus, Rivaroxaban, Argatroban, CoCr alloys, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
11. Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel or other P2Y12 inhibitors
12. Patient has severe renal dysfunction (CKD IV or V, eGFR <30) or is on dialysis
13. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
14. Patient has had a significant GI or urinary bleed within the past six months
15. Women of childbearing potential (unless they have a negative pregnancy test within 7 days of index procedure), or women who are pregnant or nursing
16. Patient has other medical conditions or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation, or be associated with a limited life expectancy (i.e., less than one year)
17. Patient is already participating in another clinical study which has not reached the primary endpoint (long-term follow-up or observational studies are permitted)

    Angiographic Exclusion Criteria
18. Patient with vessel rupture and/or visible pericardial effusion
19. Target lesion aorto-ostial location or within 5mm of the origin of the vessel (LAD, LCX, RCA)
20. Target lesion is severely calcified and/or requires use of rotational atherectomy or cutting balloon, the use of shockwave or scoring balloon is allowed
21. Target Lesion located in the Left Main artery
22. Target Lesion located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
23. Target Lesion involves a bifurcation >2.5 mm, or which requires a planned 2 or more stent technique
24. Previous placement of a stent within 10 mm of a target lesion
25. Another clinically-significant lesion (> 50%) is located in the same major epicardial vessel as a target lesion
26. Target vessel was previously treated with any type of PCI < 6 months prior to index procedure
27. Unsuccessful or complicated PCI in a non-target vessel < 48 hours prior to index procedure
28. Target vessel has a planned staged PCI ≤ 6 months after the index procedure

    Additional Exclusion Criteria for PK study:
29. Target vessel was previously treated with any type of PCI < 6 months prior to index procedure
30. Patient with planned staged PCI within 90 days after study procedure
31. Patients who have a non-target lesion treated during the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 3 days or through hospital discharge, whichever comes first
  defined as a per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target lesion revascularization

SECONDARY OUTCOMES:
Acute success | during hospital stay with a maximum of first seven days post index procedure
  defined as the successful delivery of the designated device and a final residual stenosis < 30% by QCA without TLF
Target lesion failure | 30 days
  defined as a per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target lesion revascularization
Target lesion failure | 6 months
  defined as a per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target lesion revascularization
Target lesion failure | 12 months
  defined as a per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target lesion revascularization
Target lesion failure | 2 years
  defined as a per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target lesion revascularization
Target lesion failure | 3 years
  defined as a per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target lesion revascularization
Death | 3 days or through hospital discharge, whichever comes first
  Cardiovascular and Non-cardiovascular
Death | 30 days
  Cardiovascular and Non-cardiovascular
Death | 6 months
  Cardiovascular and Non-cardiovascular
Death | 12 months
  Cardiovascular and Non-cardiovascular
Death | 2 years
  Cardiovascular and Non-cardiovascular
Death | 3 years
  Cardiovascular and Non-cardiovascular
Myocardial Infarction | 3 days or through hospital discharge, whichever comes first
  Q-wave and non-Q-wave; Target vessel and non-target vessel
Myocardial Infarction | 30 days
  Q-wave and non-Q-wave; Target vessel and non-target vessel
Myocardial Infarction | 6 months
  Q-wave and non-Q-wave; Target vessel and non-target vessel
Myocardial Infarction | 12 months
  Q-wave and non-Q-wave; Target vessel and non-target vessel
Myocardial Infarction | 2 years
  Q-wave and non-Q-wave; Target vessel and non-target vessel
Myocardial Infarction | 3 years
  Q-wave and non-Q-wave; Target vessel and non-target vessel
Target Lesion Revascularization | 3 days or through hospital discharge, whichever comes first
  Clinically indicated and non-clinically indicated
Target Lesion Revascularization | 30 days
  Clinically indicated and non-clinically indicated
Target Lesion Revascularization | 6 months
  Clinically indicated and non-clinically indicated
Target Lesion Revascularization | 12 months
  Clinically indicated and non-clinically indicated
Target Lesion Revascularization | 2 Years
  Clinically indicated and non-clinically indicated
Target Lesion Revascularization | 3 Years
  Clinically indicated and non-clinically indicated
Target Vessel Failure | 3 days or through hospital discharge, whichever comes first
  per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target vessel revascularization
Target Vessel Failure | 30 days
  per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target vessel revascularization
Target Vessel Failure | 6 months
  per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target vessel revascularization
Target Vessel Failure | 12 months
  per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target vessel revascularization
Target Vessel Failure | 2 years
  per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target vessel revascularization
Target Vessel Failure | 3 years
  per-subject composite endpoint of cardiovascular death, target vessel MI, and clinically-indicated target vessel revascularization
Late Lumen Loss | 6 months
  powered secondary endpoint assessed by QCA in a subset of patients
Optical Coherence Tomography (OCT) imaging | Post procedure and 6 months
  assessment of the lesion and stent in a subset of patients.
Pharmacokinetic profile of the drugs on the DESyne BDS Plus Stent | pre-treatment, and post-treatment at 10 minutes, 30 minutes, 1, 2, 4, 6, 12, 24, 72 hours, and 7 days
  assessment of the blood pharmacokinetics of the three drugs eluted from the DESyne BDS Plus after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, PHD, Principal Investigator — Ziekenhuis Netwerk Antwerpen (ZNA) Middelheim, Antwerp, Belgium; Mark Webster, MBChB, Principal Investigator — Auckland City Hospital
Locations (14):
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - Ziekenhuis Oost-Limburg, Campus Sint Jan, Genk
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (2):
  - Instituto Dante Pazzanese, São Paulo
  - Instituto do Coração da Faculdade, São Paulo
- General University Hospital, Prague, Czechia
- Catharina Hospital, Eindhoven, Netherlands
- New Zealand (6):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No